CLINICAL TRIAL: NCT01399892
Title: Effects of Fiber Supplementation on Glycemic Excursions and Incidence of Hypoglycemia in Children With Type 1 Diabetes
Brief Title: Effect of Fiber Supplementation in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Aida Lteif, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-002142
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: soluble fiber in the form of benefiber — Benefiber, sugar free in an amount to total 20gms/1000kcal/day of fiber

SUMMARY:
High fiber foods are recommended as a preferential source of carbohydrate by the Nutrition Study Group of the European Association for the Study of Diabetes. Dietary fibers may delay glucose absorption and reduce postprandial glycemic excursion. They also appear to have a beneficial effect on cholesterol levels. It has been shown, in few short term adult studies, that high fiber foods reduce postprandial blood glucose levels. The American Diabetes Association feels that there is little evidence confirming the positive effect of high fiber foods on blood glucose control. It is not clear whether a high fiber diet can improve glycemic control and/or reduce the risk of hypoglycemic events. Our hypothesis is that children with type 1 diabetes will benefit from having added fibers in their diet. The investigators plan to study blood glucose values using a continuous blood glucose monitor before and after dietary fibers are introduced. This will help us determine whether a diet rich in fiber should be recommended in all children with type 1 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are: Diagnosis of type I diabetes for at least two years prior to enrollment, the ability tolerate wearing the continuous blood glucose monitoring device for a total of 6 days, and the ability to follow a prescribed meal plan.

Exclusion Criteria:

* The exclusion criteria are: Medical conditions that could potentially affect the absorption of nutrients such as celiac disease of inflammatory bowel disease and the use of any fiber supplements at home.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
incidence of hypoglycemia after fiber supplementation | continuous glucose monitoring over 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aida N Lteif, MD, Principal Investigator — Mayo Clinic